CLINICAL TRIAL: NCT01475084
Title: Cryobiopsy or Forceps Biopsy During Semirigid Thoracoscopy: a Comparative Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University Clinic of Pulmonary and Allergic Diseases Golnik (Other)
Responsible Party: Principal Investigator, Aleš Rozman, MD, The University Clinic of Pulmonary and Allergic Diseases Golnik
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: Endo-0003
Record Dates: First submitted 2011-11-16; First posted 2011-11-21 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Pleural Effusion; Pleural Diseases
Keywords: Flex-rigid pleuroscopy; cryobiopsy; pleural biopsy; pleural effusion; safety; thoracoscopy
MeSH Terms: conditions — Pleural Effusion; Pleural Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cryobiopsy, forceps biopsy (Experimental): Cryoiopsies will be obtained by flexible autoclavable cryoprobe 20416-032 (Erbokryo CA, ERBE, Germany) with 2.4 mm in diameter. The tip of the probe is cooled to -890C with nitrous oxide within seconds after footswitch activation.
  Forceps biopsies will be obtained by flexible FB-55CD-1 Olympus forceps.
  Interventions: Device: cryobiopsy (Autoclavable cryoprobe 20416-032 (ERBE, Germany) Flexible FB-55CD-1 Olympus forceps

INTERVENTIONS:
Device: cryobiopsy (Autoclavable cryoprobe 20416-032 (ERBE, Germany) Flexible FB-55CD-1 Olympus forceps — The tip of the cryoprobe will be attached to suspicious part of parietal pleura and activated by footswitch for 3 seconds. The frozen tissue is going to be extracted by gently pulling of the probe. The probe with the attached biopsy sample is going to be removed together with the thoracoscope through trocar. The biopsy sample will be released from the probe by thawing in the saline.
  Forceps biopsy will be performed on usual way.
  Other Names: Autoclavable cryoprobe 20416-032 (ERBE, Germany); Flexible FB-55CD-1 Olympus forceps

SUMMARY:
The purpose of this study is to compare cryobiopsies with forceps biopsies during semirigid thoracoscopy.

DETAILED DESCRIPTION:
The investigators are going to compare diagnostic yield and size, morphological features, immunohistochemistry as measures of the quality of the samples. The secondary aim is to evaluate safety with focus on bleeding intensity.

ELIGIBILITY:
Inclusion Criteria:

* 18 or more years old
* unilateral pleural effusion of unknown origin
* pleural irregularities suspicious for pleural malignancy
* referral for thoracoscopy after less invasive means of diagnosis had failed

Exclusion Criteria:

* uncontrolled bleeding tendency
* unstable cardiovascular status
* severe heart failure
* ECOG performance status 4
* persistent hypoxemia after evacuation of pleural fluid
* pleural symphisis, fibrothorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Comparison of forceps biopsy and cryobiopsy samples | 12 month
  * diagnostic yield
  * size of the biopsy specimens in mm2
  * interpretability of biopsy specimens in histopathology terms: 1. easily interpretable (enough tissue with all elements required for diagnosis) 2. interpretable with some difficulty (less tissue or diagnostic elements - diagnosis less reliable) 3. interpretable with great difficulty (little tissue or scarce diagnostic elements - low reliability of diagnosis) 4. non-interpretable (diagnosis not possible)
  * assessment of biopsy-related artifacts by describing the amount of unaltered tissue in quartiles

SECONDARY OUTCOMES:
Safety | 1 month
  The degree of bleeding at the biopsy site will be assessed as 1 = slight, self-limited, 2 = moderate, requiring electrocautery intervention, 3 = severe, requiring interruption of the procedure, chest tube drainage and intravenous fluid resusucitation.

CONTACTS AND LOCATIONS:
Overall Officials: Ales Rozman, MD, Principal Investigator — University Clinic Golnik
Locations (1):
- University Clinic Golnik, Golnik, Golnik, Slovenia